CLINICAL TRIAL: NCT05994274
Title: A Prospective Clinical Study of Association Between Postoperative Dyslipidemia and Organ
Brief Title: A Clinical Study of Association Between Postoperative Dyslipidemia and Organ Rejection in Transplant Patients
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: WuhanUH-XJH
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Heart Transplant Failure and Rejection
Keywords: heart transplantation; Macrophages; Fatty acid; PCSK9; Lipid metabolism
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HTx: Patients after heart transplantation.

SUMMARY:
Abnormal lipid metabolism is a common complication after organ transplantation, with pathological changes in lipid parameters occurring in approximately 60-80% of cardiac transplant recipients receiving triple immunotherapy with cyclosporine, imid azathioprine, and methylprednisolone. With the significant increase in long-term survival and increasing age of transplant patients, atherosclerotic cardiovascular diseases, such as those caused by dyslipidemia, have become a major cause of transplant organ failure and recipient death. However, the causes of dyslipidemia after organ transplantation, as well as the effects and mechanisms of dyslipidemia on transplant rejection, are unknown.

Previous studies have found that 1. increased lipid levels occur in recipients after heart transplantation; 2. during rejection, hepatic PCSK9 expression is increased in recipients; 3. a high-fat environment increases the immunoreactivity of human peripheral blood lymphocytes. It is suggested that PCSK9-lipid disorder-immune cell interactions may be associated with the development of transplant rejection.

In this project, we propose to (1) establish a long-term follow-up system for postoperative cardiac transplantation patients in our department to track the characteristics of lipid changes in transplantation patients, to clarify the link between dyslipidemia and rejection, and to provide a strong evidence-based medical basis for the management of lipids during the perioperative period and in the postoperative period; (2) expand the dimensions of lipid-related assays under the support of the above system, and to incorporate transcriptomic, proteomic, and metabolomic research methods to elucidate transplantation rejection in a multidimensional manner. (ii) Expanding the dimensions of lipid-related assays to include transcriptomic, proteomic, and metabolomic studies to elucidate the relationship between PCSK9 and dyslipidemia in transplant patients; (iii) Adopting single-cell sequencing technology to deeply reveal the potential mechanism by which changes in lipids affect T-cell-mediated rejection of cardiac transplants. The mechanism of T-cell-mediated cardiac transplantation rejection is revealed by single-cell sequencing.

ELIGIBILITY:
Inclusion Criteria:

* After heart transplantation
* Age ≥ 18
* Disease duration: symptomatic heart failure ≥ 6 months prior to screening date
* The patient's informed consent

Exclusion Criteria:

* Refusal of the patient to provide consent
* Suspected poor capability to follow instructions and cooperate
* Another life-threatening disease with poor prognosis (survival less than 2 years)
* Participation in any other clinical study within less than 30 days prior to screening date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone heart transplant.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Blood lipid measurements | 4 years
  TG, TC, HDL-C, LDL-C, ApoB
Graft/Patient survival | 4 years

SECONDARY OUTCOMES:
Left ventricular ejection fraction (LVEF) at rest | 4 years
  determined by contrast echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, China

IPD SHARING:
Plan to Share IPD: No